CLINICAL TRIAL: NCT03849053
Title: The Effectiveness of Mézières Therapy in the UCAM's Athletes With Low Back Pain
Brief Title: Mézières Therapy in the UCAM's Athletes With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Orges Lena, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB8334280
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain; Postural; Strain
Keywords: Low back pain; Mézières method; Postural treatment; Athletes
MeSH Terms: conditions — Low Back Pain; Sprains and Strains

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mézières method (Experimental)
  Interventions: Other: Mézières Therapy for Low back pain
- Control Group (Active Comparator)
  Interventions: Other: Mézières Therapy for Low back pain

INTERVENTIONS:
Other: Mézières Therapy for Low back pain — Spinal muscular global stretching

SUMMARY:
The purpose of this research study focuses on the re-harmonization of the kinetic chains and posture based on spinal muscular atrophy and global stretching while trying to test the effectiveness of Mézières therapy on sports subjects with low back pain.

DETAILED DESCRIPTION:
The experimental study was conducted on 139 young athletes of National Rhythmic Gymnastics of Murcia, UCAM Murcia CF and UCAM Murcia CB/EBA during a six months period in the city of Murcia. Precisely, the Mézières therapy was conducted in an experimental group of 69 athletes and in a control group with other 70 athletes with Low Back Pain. This study is developed through a cycle of global stretching decompensate interventions on the athletes with postural alterations and vertebral pain at 95% confidence level. The statistical analysis was handled by using the univariate general linear model with the support of SPSS statistics.

ELIGIBILITY:
Inclusion Criteria:

* between 15 - 39 years
* athletes with low back pain lasting more than 1 month
* scoliosis
* kyphosis

Exclusion Criteria:

* presence of tumors or spinal metastases
* vertebral fractures
* osteoporosis
* infection or inflammation in acute diseases with involvement of the central nervous system
* herniated discs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
VAS (Visual Analogic Scale) | 6 months
  It consists in identifying the patient, on a 10 cm line, the point that best represents his pain, where 0 means no pain and 10 = worst possible pain.
Sit and Reach flexibility test | 6 months
  Designed to test the flexibility of lower back and hamstring muscles and is important as a result of lumbar lordosis, forward pelvic tilt and lower back pain. The score is recorded to the nearest inch/cm or inch/cm as the distance reached by the hand. For women, the lowest value is ˂ -15 cm and the highest is ˃ +30 cm. For men instead, the lowest value is ˂ -20 cm and the highest is >+27 cm.
Runtastic Performance Pedometer | 6 months
  - Runtastic PRO is an app aimed at recording fitness in many activities and sports. It captures all basic data: distance, average speed, speed between mile markers, altitude, pace, step between mile markers, duration, calories burned and route plotted on a map using Global Positioning System. The final result shows how many steps are made in the arc of the minute (st / 60sec).

SECONDARY OUTCOMES:
Roland-Morris Questionnaire (CRM) | 6 months
  Measures the physical disability of athletes and consists of 24 points of functional capacity of the back. The sense of progression is: the more serious the worse is the performance.
Health status questionnaire (SF-12) | 6 months
  The questionnaire consists in 12 items of the 8 dimensions of the SF-36 (124) such as: physical function (2), social function (1), physical role (2), emotional role (2), mental health (2), vitality (1), body pain (1), general health (1). Meanwhile response options forms Likert-type scales that evaluate intensity or frequency are achieved.